CLINICAL TRIAL: NCT01391520
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Deferiprone in the Reduction of Morbidity and Mortality in Patients With Chronic Kidney Disease Undergoing Diagnostic or Interventional Cardiac Procedures and Receiving an Iodinated Radiocontrast Agent
Brief Title: Efficacy and Safety of Deferiprone in Patients With Chronic Kidney Disease Undergoing a Cardiac Catheterization and Receiving Contrast Agent
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor encountered funding issues for this study.
Sponsor: CorMedix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRMD001-3001
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Contrast-Induced Nephropathy; Labile Iron; Iron Chelation; Deferiprone
MeSH Terms: conditions — Acute Kidney Injury | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CRMD001-Deferiprone (Experimental): CRMD001 represents unique formulations of Deferiprone. Subjects will be given one (900 mg) immediate release and two (900 mg) extended release tablets 1-3 hours prior to angiography and then every 12 hours for a total of 8 days
  Interventions: Drug: deferiprone
- Placebo (Placebo Comparator): 3 placebo tablets matching the appearance of the experimental treatment arm (CRMD001) will be given every 12 hours for a total of 8 days, beginning 1-3 hours prior to angiography
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: deferiprone — 3 tablets (treatment arm assigned in double-blind, randomized manner) will be given every 12 hours for a total of 8 days, beginning 1-3 hours prior to angiography
  Arms: CRMD001-Deferiprone
Drug: Placebo — 3 tablets (treatment arm assigned in double-blind, randomized manner) will be given every 12 hours for a total of 8 days, beginning 1-3 hours prior to angiography
  Arms: Placebo

SUMMARY:
This trial will evaluate whether treatment with CRMD001 (unique formulations of the iron chelator, Deferiprone) will reduce morbidity and mortality in subjects with Chronic Kidney Disease (CKD) and additional risk factors. Adult subjects with moderate to severe CKD who are undergoing diagnostic or interventional coronary angiography will be randomized to either placebo or CRMD001 and followed for 90 days. Subjects will receive 8 days of randomized therapy starting 1-3 hours prior to angiography. The primary endpoint of the trial will be the difference in a composite of specified renal and cardiovascular clinical events occurring through Day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. eGFR between 15 ml/min/1.73 m2 and < 60 ml/min/1.73 m2
3. Presence of at least one additional risk factor:

   * Diabetes Mellitus type 1 or 2
   * Age ≥ 75 years
   * Left Ventricular Ejection Fraction ≤ 40%

Exclusion Criteria:

1. End-Stage Renal Disease
2. Primary PCI for STEMI
3. Currently receiving mechanical ventilation
4. Known active liver disease or liver failure
5. Evidence of hemodynamic instability, such as a requirement for pressor agents
6. Exposure to contrast media within prior 10 days
7. Currently receiving fenoldopam, dopamine, theophylline, aminophylline, mannitol, or Ascorbic acid (> 2 g/day)
8. Absolute neutrophil count < 1500

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Estimated); Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
A composite of renal and cardiovascular clinical events occurring through Day 90 | Day 90 following index cardiac catheterization